CLINICAL TRIAL: NCT04488939
Title: A Prospective, Open-label Evaluation of Restylane® Skinboosters™ Vital in the décolletage Region
Brief Title: Restylane® Skinboosters™ Vital in the décolletage Region
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-Gal-SBV
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2020-07

CONDITIONS: Decolletage Rejuvenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bilateral treatment (Experimental)
  Interventions: Device: Restylane® Skinboosters™ Vital (SBV)

INTERVENTIONS:
Device: Restylane® Skinboosters™ Vital (SBV) — Hyaluronic acid

SUMMARY:
Restylane® Skinboosters™ Vital (SBV) is a smooth formulation without particles, which helps it distribute evenly and smoothly under the skin to aid in rejuvenation. This feature makes RSV particularly well suited for more superficial injections, such as at the level of the dermis.

SBV smooths fine lines and wrinkles and is intended to improve skin smoothness and appearance, as well as the elasticity and hydration of the skin in the face and dorsal hands. However, many clinicians have used SBV in other regions of the body. Given these attributes, SBV are particularly well suited for photo aged skin. A region that is susceptible to photo-ageing and may therefore benefit from the use of SBV is the décolletage. Photodamaged skin of the chest is characterized by atrophy, skin laxity, fine lines and wrinkles, dehydration and tactile roughness. Therefore, SBV may help to improve these signs of aging in the décolletage region.

Study Aim: To investigate the effectiveness and tolerability of SBV for rejuvenation of the décolletage region.

ELIGIBILITY:
Inclusion Criteria:

1. A score > 2 on the GDS, as assessed by the treating physician at Baseline.
2. Females aged > 25 and < 70
3. Ability to adequately understand the verbal explanations and the written subject information provided in local language and ability and willingness to give consent to participate in the study.
4. Signed and dated informed consent to participate in the study and unrestricted use of décolletage images for marketing purpose.
5. If female of childbearing potential: a negative urine pregnancy test before all treatments is required.

Exclusion Criteria:

1. Current Pregnancy or lactation [sexually active women of childbearing age must agree to use medically acceptable methods of contraception for the duration of this study (e.g., oral contraceptives, condoms, intrauterine device, shot/injection, patch)];
2. Patients meeting any official Restylane contra-indications;
3. Inability to comply with follow-up and abstain from other treatments in the region of interest during the study period;
4. Heavy smokers, classified as smoking more than 12 cigarettes per day;
5. History of severe or multiple allergies manifested by anaphylaxis;
6. Previous tissue revitalization therapy in the treatment area within 6 months before treatment with laser or light, mesotherapy, radiofrequency, ultrasound, cryotherapy, chemical peeling, or dermabrasion;
7. Subjects presenting with known allergy to hyaluronic acid (HA) filler or amide local anesthetics.
8. Subjects presenting with porphyria.
9. Subjects with active disease, such as inflammation, infection or tumors, in or near the intended treatment site.
10. Subjects with bleeding disorders or in subjects who are taking thrombolytics or anticoagulants.
11. Subjects using immunosuppressants.
12. History of other décolletage treatment/procedure in the previous 6 months below the level of the neck that, in the treating investigator's opinion, would interfere with the study injections and/or study assessments or exposes the subject to undue risk by study participation.
13. Tattoos, piercings or visible markings that in the treating investigator's opinion, may interfere with results or assessments [excessive sun damage, tan lines, dark spots, moles, scars (hypertrophic, keloid), tan lines].
14. Cancer or precancer in the treatment area, e.g. actinic keratosis;
15. History of bleeding disorders or treatment with thrombolytics, anticoagulants, or inhibitors of platelet aggregation (e.g. Aspirin or other non-steroid anti-inflammatory drugs [NSAIDs]), within 2 weeks before treatment;
16. Patients using immunosuppressants;
17. Patients with a tendency to form hypertrophic scars or any other healing disorders;
18. Patients with known hypersensitivity to lidocaine or agents structurally related to amide type local anesthetics (e.g., certain anti-arrhythmics);
19. Patients with epilepsy, impaired cardiac conduction, severely impaired hepatic function or severe renal dysfunction.

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Galderma Décolletage Scale | Visit 4, Week 12
  Proportion of subjects achieving at least a one-point improvement on the Galderma Décolletage Scale (GDS), one month following the treatment regime (i.e., Visit 4; Week 12; one month after completing three treatments, each spaced one month apart). Scores: 0 (none) to 4 (severe)

SECONDARY OUTCOMES:
Galderma Décolletage Scale | Visit 5 and 6 (Weeks 16 and 20)
  Proportion of subjects achieving at least a one-point improvement on the Galderma Décolletage Scale , at Visits 5 and 6 (i.e., 2- and 3-months post treatment regime). Scores: 0 (non) to 4 (severe)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, FRCSC, Principal Investigator — Erevna Innovations Inc.
Locations (1):
- Erevna Innovations Inc, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No